CLINICAL TRIAL: NCT01070732
Title: An Open-label Non-randomized Phase IV Trial of the Clinical Efficacy of Intravenously Administered 1000mg Paracetamol as Antipyretic and Analgesic Medication
Brief Title: Paracetamol as Antipyretic and Analgesic Medication
Acronym: APOTEL01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Evangelos Giamarellos-Bourboulis, Assistant Professor of Medicine, University of Athens, Medical School
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APOTEL01
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Fever; Analgesia
Keywords: Fever; Infectious diseases; Neoplasia; Pain; cholecystectomy; Colectomy
MeSH Terms: conditions — Fever; Agnosia; Communicable Diseases; Neoplasms; Pain | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paracetamol (Experimental): All patients will receive one single dose of 1000mg paracetamol.
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — All patients will receive one single dose of 1000mg paracetamol. If considered mandatory by the attending physician, similar doses may be administered latter for a maximum period of five days. The maximum allowed daily dose is 3000mg. If the attending physician believes that after the administration of at least of three doses the desired analgesic or antipyretic effect is not achieved, he may administer any other compound in his will.
  Other Names: ΑPOTEL®

SUMMARY:
The present study is aiming to unravel the clinical efficacy of intravenously administered paracetamol as antipyretic and analgesic medication in various medical conditions.

DETAILED DESCRIPTION:
Although modern therapeutics is targeting at prolongation of survival, despite the underlying illness, it also aims at the improvement of the quality of life. Two major symptoms affect considerably quality of life, fever and pain. Both symptoms are common denominators of a vast number of clinical situations some of which have good prognosis and some of which do not have. Among them situations like infectious diseases, hematologic malignancies, solid tumor malignancies, connective tissue disorders and factors connected to surgical operations predominate. Post-operative pain extents too long and imposes severely on the post-operative course of the patient.

A variety of compounds have been developed for the management of fever and pain, the most successful being non-steroidal anti-inflammatory drugs. They exist in a variety of forms for various types of administration. Those administered parenterally are considered more efficacious than those administered orally in terms of the rate of the achieved clinical effect. Furthermore, several conditions necessitate parenteral administration.

Paracetamol is a well-known antipyretic and analgesic compound available for many years for oral administration since intravenous infusion was hampered by water insolubility. Its pro-drug, namely, pro-paracetamol, was applied for intravenous infusion where an amount of 2g was equally potent to 1 g of paracetamol. Pro-paracetamol has been given with success as analgesic medication in women undergoing laparoscopic operation, as antipyretic in patients with hematologic malignancies, as antipyretic in children bearing infectious diseases and as antipyretic in critically ill patients.

Ready-made paracetamol for intravenous infusion has been in the market in some European countries. It has been tested in four clinical trials. In the first trial it was given as post-operative analgesia at a dose of 1g x 4 in 80 patients undergoing laparoscopic cholecystectomy. Clinical efficacy was comparable to parecoxib and valdecoxib. In three other studies, it was given as post-operative analgesia after spinal body ectomy and after resection of the third mole providing conflicting results. However, in all the three latter studies, the number of patients given paracetamol was limited.

In Greece, paracetamol for intravenous infusion at vials of 1g/6.7ml is manufactured by the company Uni-Pharma (ΑPOTEL®). Based on: a) the limited number of patients enrolled in the studies mentioned earlier, and b) the application of that form only after laparoscopic cholecystectomy and spinal body ectomy, the present study is aiming to unravel the clinical efficacy of the above formula of 1g intravenous paracetamol as antipyretic and analgesic medication in various medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Written informed consent by the patients
* Medical condition necessitating the administration of antipyretic or analgesic medications

Exclusion Criteria:

* Αge lower than 18 years
* Lack of informed consent
* History of liver cirrhosis
* Blood creatinine greater than 3mg/dl
* Blood AST greater than 3 times the upper normal level according to the lab of the participating hospital
* History of hypersensitivity to non-steroidal ant-inflammatory drugs
* History of abuse of analgesics
* Pregnancy or lactation
* Fulminant hemorrhage of the upper or lower digestive tract
* Thrombocytopenia defined as less than 50000 platelets/μl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of intravenously administered 1000mg ΑPOTEL® as antipyretic and analgesic medication. | One year

SECONDARY OUTCOMES:
Pharmacokinetics of paracetamol after intravenous infusion. | One year
Effect of paracetamol after intravenous infusion in serum inflammatory mediators | One year

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos J Giamarellos-Bourboulis, MD, PhD, Study Chair — University of Athens, Medical School; Helen Giamarellou, MD, PhD, Principal Investigator — ATTIKON University Hospital of Athens; George Koratzanis, MD, PhD, Principal Investigator — Sismanogelion General Hospital, Athens; Konstantinos Atmatzidis, MD, PhD, Principal Investigator — G.Gennimatas General Hospital of Thessaloniki
Locations (3):
- Greece (3):
  - 4th Department of Internal Medicine, ATTIKON University Hospital, Athens
  - 2nd Department of Medicine, Sismanogleion General Hospital, Athens
  - 2nd Department of Surgery, G. Gennimatas General Hospital, Thessaloniki

REFERENCES:
- [Background] Tiippana E, Bachmann M, Kalso E, Pere P. Effect of paracetamol and coxib with or without dexamethasone after laparoscopic cholecystectomy. Acta Anaesthesiol Scand. 2008 May;52(5):673-80. doi: 10.1111/j.1399-6576.2008.01650.x. PMID 18419721
- [Background] Cakan T, Inan N, Culhaoglu S, Bakkal K, Basar H. Intravenous paracetamol improves the quality of postoperative analgesia but does not decrease narcotic requirements. J Neurosurg Anesthesiol. 2008 Jul;20(3):169-73. doi: 10.1097/ANA.0b013e3181705cfb. PMID 18580346
- [Background] Grundmann U, Wornle C, Biedler A, Kreuer S, Wrobel M, Wilhelm W. The efficacy of the non-opioid analgesics parecoxib, paracetamol and metamizol for postoperative pain relief after lumbar microdiscectomy. Anesth Analg. 2006 Jul;103(1):217-22, table of contents. doi: 10.1213/01.ane.0000221438.08990.06. PMID 16790656